CLINICAL TRIAL: NCT04512963
Title: A Phase I, Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose (SAD) Study Including a Food Interaction Study, Followed by a Multiple Ascending Dose (MAD) Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamic Profile of Progerinin in Healthy Volunteers
Brief Title: Phase I Study of Progerinin in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PRG Science & Technology Co., Ltd. (Industry)
Collaborators: Amarex Clinical Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRG-PRO-001
Record Dates: First submitted 2020-08-06; First posted 2020-08-14 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Hutchinson-Gilford Progeria Syndrome; Werner Syndrome
Keywords: HGPS; WS; Progeria
MeSH Terms: conditions — Progeria; Werner Syndrome

STUDY DESIGN:
Intervention Model Description: SAD Phase including Food Interaction:
  This is a randomized, double-blind, placebo-controlled, dose-escalating study in healthy volunteers. Participants will be assigned to 1 of up to 6 cohorts and will be randomized within each cohort to Progerinin or placebo at 3:1 ratio.
  Following the completion of the SAD phase, if study stopping criteria (SSC) is not met, then participants in cohort 5 and 6 will cross-over to the fed part of the study following a 7 day washout period. If SSC is achieved in the SAD phase, then the previous dose will be in the Food Interaction phase.
  MAD Phase:
  This is a randomized, double-blind, placebo-controlled, dose-escalating study in healthy volunteers. If SSC is not met in the SAD phase, then participants will be assigned to 1 of 2 cohorts and will be randomized within each cohort to Progerinin or placebo at 3:1 ratio. If SSC is achieved in the SAD phase, then the previous two doses will be used as the 2 cohorts in the MAD phase.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SAD Phase including Food Interaction (Experimental): Single Ascending Dose (SAD) study with up to 6 cohorts + Food interaction phase on two cohorts
  Interventions: Drug: Progerinin; Drug: Placebo
- MAD Phase (Experimental): Multiple Ascending Dose (MAD) study with up to 2 cohorts
  Interventions: Drug: Progerinin; Drug: Placebo

INTERVENTIONS:
Drug: Progerinin — 100 mg/g nano-suspension for oral use
  Other Names: SLC-D011
Drug: Placebo — A substance that has no therapeutic effect, used as a control in testing Progerinin
  Other Names: Vehicle control

SUMMARY:
PRG-PRO-001 is a Phase I, Randomized, Double-blind, Placebo-Controlled, Single Ascending Dose (SAD) Study including a food interaction study, followed by a Multiple Ascending Dose (MAD) Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamic Profile of Progerinin in Healthy Volunteers. This is a first-in-human study. The study aims to determine the safety and tolerability of Progerinin after single and multiple doses in healthy volunteers and to evaluate the pharmacokinetics (PK) of Progerinin after single and multiple dose administrations in healthy volunteers.

DETAILED DESCRIPTION:
PRG Science & Technology Co., Ltd. (PRG S&T) is developing Progerinin (SLC-D011) for the treatment of the rare aging diseases Hutchinson-Gilford Progeria Syndrome (HGPS) and Werner Syndrome (WS).

Progerin, an abnormal splice variant of the inner nuclear membrane protein lamin A is implicated in the pathology of HGPS and WS. It is believed that the extremely strong binding between lamin A and progerin is responsible for the nuclear abnormality phenotype observed in HGPS. WS is caused by functional defect of WRN, RecQ4L DNA helicase and rapid accumulation of progerin in WRN deficient condition is thought to be the cause of premature aging in WS. PRG S&T has shown that Progerinin binds specifically to progerin reduces its expression in both HGPS and WS cells, Progerinin further prevents progerin-lamin A in HGPS cells. In a progeria mouse model (LmnaG609G/G609G), treatment with Progerinin via intraperitoneal (i.p) injection (20 mg/kg, twice per week) could increase the body weight and extend the life span of LmnaG609G/G609G mice up to 21 weeks. In the LmnaG609G/+ mouse model, improved morphology such as status of coat hair and body size, increased body weight and extended life span for about 16 weeks was noted following Progerinin treatment. In addition, Progerinin can suppress muscle weakness including the heart muscle. Safety pharmacology studies did not indicate any Progerinin-related effects on vital organs and systems including respiratory, cardiovascular and central nervous system.

Prior to studies in the disease states, this study PRG-PRO-001, an initial first-in-human study, will be conducted in healthy volunteers to assess the safety, tolerability and pharmacokinetics of Progerinin. PRG-PRO-001 is a Phase I, Randomized, Double-blind, Placebo-Controlled, Single Ascending Dose (SAD) Study including a food interaction study, followed by a Multiple Ascending Dose (MAD) Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamic Profile of Progerinin in Healthy Volunteers. This is a first-in-human study. The study aims to determine the safety and tolerability of Progerinin after single and multiple doses in healthy volunteers and to evaluate the pharmacokinetics (PK) of Progerinin after single and multiple dose administrations in healthy volunteers. The estimated enrollment is around 56 healthy volunteers, with 40 subjects estimated for the SAD phase and 16 subjects for the MAD Phase at one site in the USA.

Expanded Access Program is available. For more details, please use the link in the References Section below to access our company's main webpage on Expanded Access Program.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be eligible for enrollment in the study only if they meet ALL of the following criteria:

1. Healthy male and female subjects, 18 to 45 years of age, inclusive.
2. The subject has a body mass index (BMI) of 18.0 to 30.0 kg/m2, inclusive, and weighs at least 50 kg.
3. The subject is in good health and has no medical condition of clinical significance or that may impact the outcome of the study, as determined by the investigator (as determined by medical history, physical examination, 12-lead electrocardiogram [ECG], vital signs, and clinical laboratory results at screening).
4. The subject is able to understand the nature of the study and any potential hazards associated with participating in it.
5. The subject is able to communicate satisfactorily with the investigator and to participate in, and comply with, the requirements of the study.
6. The subject is willing to provide written informed consent to participate in the study after reading the informed consent form and the information provided, and has had the opportunity to discuss the study with the investigator or designee.
7. Negative pregnancy test for female subjects. Women of child bearing potential (WOCBP) and Women not of child bearing potential are eligible to participate. Both women of child bearing potential and women of no child bearing potential should use an approved method of birth control and agrees to continue to use this method for the duration of the study (and for 90 days after taking the last dose of Progerinin).

   Acceptable methods of contraception include abstinence, female subject/partner's use of hormonal contraceptive (oral, implanted, or injected) in conjunction with a barrier method (WOCBP only), female subject/partner's use of an intrauterine device (IUD), or if the female subject/partner is surgically sterile or 2 years post-menopausal. All male subjects/partners must agree to consistently and correctly use a condom for the duration of the study and for 90 days after taking the study drug. In addition, subjects may not donate sperm for the duration of the study and for 90 days after taking study drug.
8. Subjects not taking any medications or dietary supplements (i.e., St. John's Wort and goldenseal) which are inhibitors or inducers of CYP 3A4 and CYP 2D6 during screening and for the duration of the trial.
9. Subjects not taking any medications which are substrates of CYP2C8, CYP2C9, CYP2C19, CYP2D6, CYP3A4/5 during screening and for the duration of the trial.

Exclusion Criteria:

Subjects will be eligible for enrollment in the study only if they meet NONE of the following criteria:

1. The subject has a history of severe allergic or anaphylactic reactions.
2. The subject has a known allergy or hypersensitivity to any component of the formulation.
3. The subject has a medical history or current evidence of any clinically significant (as determined by the investigator) cardiac, endocrine (including diabetes), hematologic, hepatobiliary (abnormal 12lanine aminotransferase [ALT], aspartate aminotransferase [AST], gamma-glutamyl transpeptidase [GGT], or total bilirubin), immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, or renal condition, or other major disease.
4. The subject has a history of any malignant disease.
5. The subject has a history of more than one herpes zoster episode or multimetameric herpes zoster.
6. The subject has a history of an opportunistic infection (e.g. cytomegalovirus, pneumocystis carinii, aspergillosis, clostridium difficile).
7. The subject has a history of or ongoing chronic or recurrent infectious disease (e.g. infected indwelling prosthesis, osteomyelitis, chronic sinusitis).
8. The subject has had major trauma or surgery in the 2 months before screening or at any time between screening and check-in.
9. The subject has had an acute infection within 2 weeks before screening or at any time between screening and check-in including, but not limited to, history, signs, or symptoms of a common cold (eg, mild rhinorrhea), untreated oral/dental abnormalities (e.g. untreated dental caries as determined by examination of the mouth), or untreated disruption of the skin.
10. The subject has clinically significant abnormal ECG findings at screening, check-in visits, or predose, as determined by the Investigator.
11. The subject has a supine blood pressure measurement outside the ranges of 90 to 140 mm Hg systolic or 45 to 90 mm Hg diastolic (measured after a rest of at least 5 minutes) at screening, check-in, or predose. Note: If either value is out of the range, blood pressure measurements may be repeated in the supine position at intervals of 5 to 10 minutes up to 3 times. If the mean systolic or diastolic measurement continues to exceed the stated limits, the subject will be excluded.
12. The subject has a pulse of fewer than 45 beats per minute (bpm) or greater than 100 bpm (measured after a rest of at least 5 minutes) at screening, check-in, or predose.
13. The subject tests positive for tuberculosis (TB) at screening by the QuantiFERON-TB Gold Test, or has a history of latent, inadequately treated, or active TB.
14. The subject has a known history of, or a positive test result for, hepatitis B surface antigen (HbsAg), hepatitis C virus (HCV), or human immunodeficiency virus (HIV) types 1 or 2 at screening.
15. The subject has used prescription or over-the-counter (OTC) medication (other than ≤2 g/day paracetamol [acetaminophen] or ≤800 mg/day ibuprofen), vitamins, or herbal remedies, within 2 weeks or 5 half-lives before study drug administration, whichever is longer.
16. The subject has participated in another clinical study of a new investigational drug or has received an investigational drug within the 3 months or 5 half-lives (if available) before study drug administration, whichever is longer.
17. The subject has had a loss of more than 400 mL of blood (e.g. a blood donation) within 2 months before study drug administration, or has received any blood, plasma, or platelet transfusions within 3 months before check-in, or plans to donate blood during the study or within 3 months after the study.
18. The subject has a history of alcohol abuse (defined as an alcohol intake more than 21 units per week) or a history of drug abuse within the 6 months before study drug administration, or a history of substance abuse deemed significant by the investigator. A unit of alcohol is defined as 240 mL of beer, 120 mL of wine, or 1 single shot of spirits. The subject will be required to abstain from alcohol consumption 48 hours prior to screening or check-in.
19. The subject is a current smoker or has a history of smoking.
20. The subject has a positive test for alcohol or drugs of abuse (barbiturates, methamphetamine, benzodiazepines, morphine/opiates, phencyclidine (PCP), amphetamines, tetrahydrocannabinol (THC), methylenedioxymethamphetamine (MDMA), cocaine, methadone, and cotinine) at screening or check-in.
21. The subject is unable to participate in, or successfully complete, the study, in the opinion of their general practitioner or the investigator, because the subject is any of the following:

    1. mentally or legally incapacitated, or unable to give consent for any reason
    2. in custody due to an administrative or a legal decision, or under tutelage, or being admitted to a sanitarium or social institution
    3. unable to be contacted in case of emergency
    4. unlikely to cooperate or comply with the clinical study protocol or is unsuitable for any other reason

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2020-08-24 (Actual); Primary Completion 2021-07-27 (Actual); Study Completion 2021-07-27 (Actual)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicities (DLTs) | Day 1 through 7 days after the last study drug administration
  Any clinically significant adverse event (AE)/serious adverse event (SAE) or clinically significant laboratory abnormality which is classified as > Grade 2 (according to the National Cancer Institute Common Terminology Criteria for Adverse Events [CTCAE] version 5.0), where applicable, deemed by the investigator as at least "possibly, probably or definitely related" to Progerinin but unrelated to concurrent illness, or concomitant medications.
Incidence of Treatment-Emergent Adverse Events (TEAEs) | Day 1 through 7 days after the last study drug administration
  An adverse event (AE) is defined as any unfavorable or unintended sign, symptom, or disease that occurs or is reported by the patient to have occurred, or a worsening of a pre-existing condition. An adverse event may or may not be related to the study treatment.
Incidence of withdrawals due to Adverse Events (AEs) | Day 1 through 7 days after the last study drug administration
  Incidence of withdrawals due to Adverse Events (AEs) defined above
Incidence of abnormal blood work tests results, abnormal Urinalysis and positive Pregnancy test | At baseline, 72 to 96 hours after the last study drug administration, and on Day 7 after the first and the last study drug administration
Change in vital signs | At pre-dose, over 96 hours after study drug administration, and on Day 7 after the last study drug administration
  Vital signs measurement includes blood pressure (both systolic and diastolic blood pressures), pulse, temperature and respiratory rate.
Incidence of abnormal ECG parameters | At pre-dose, over 96 hours after study drug administration, and on Day 7 after the last study drug administration
Incidence of abnormal physical examination findings | At baseline, 96 hours after the last study drug administration, and on Day 7 after the last study drug administration
Maximum observed plasma drug concentration (Cmax) | 0-96 hours
Apparent terminal elimination half-life (t1/2) | 0-96 hours
Time to maximum observed plasma drug concentration (Tmax) | 0-96 hours
Area under the plasma drug concentration-time curve (AUC) | 0-96 hours
Percentage of AUC0-∞ extrapolated from Tlast to infinity (AUCext) | 0-96 hours
Apparent plasma clearance (CL/F) | 0-96 hours
Apparent Volume of distribution (Vz/F) | 0-96 hours

CONTACTS AND LOCATIONS:
Locations (1):
- PRG S&T Investigational Site, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: PRG S&T Expanded Access Program — http://prgst.com/bbs/board.php?bo_table=notice_eng&wr_id=6